CLINICAL TRIAL: NCT05427955
Title: Comparison of the Efficiency of Bi-Level ESPB and Single-Level ESPB for Postoperative Analgesia in Patients Undergoing VATS
Brief Title: Efficacy of Bi-level ESPB Application in Patients Undergoing VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E.Kurul-E1-22-2534
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative; Thoracic Surgery, Video-Assisted; Erector Spinae Plane Block; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-level Erector Spinae Plane Block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T5 spinous process, 30 ml of 0.25% bupivacaine hydrochloride will be injected cauda-cranially into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: One-level Erector Spinae Plane Block
- Bi-level Erector Spinae Plane Block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T4 spinous process, 15 ml of 0.25% bupivacaine hydrochloride will be injected cauda-cranially into the interfacial space below the erector spinae muscle, above the transverse process. Next, the needle will be withdrawn till subcutaneously and the linear US probe will be placed 2-3 cm lateral to the T6 spinous process. Finally, 15 ml of 0.25% bupivacaine hydrochloride will be injected cranio-caudally into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: Bi-level Erector Spinae Plane Block

INTERVENTIONS:
Procedure: One-level Erector Spinae Plane Block — One-level Erector Spinae Plane Block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, and when the patient is placed in the lateral decubitus position. In applications, 30 ml of 0.25% bupivacaine will be injected at the T5 level.
  Arms: One-level Erector Spinae Plane Block
Procedure: Bi-level Erector Spinae Plane Block — Bi-level Erector Spinae Plane Block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, and when the patient is placed in the lateral decubitus position. In applications, 15 ml of 0.25% bupivacaine at T4 level and 15 ml of 0.25% bupivacaine at T6 level will be injected.
  Arms: Bi-level Erector Spinae Plane Block

SUMMARY:
Video-assisted thoracic surgery (VATS) has become a common procedure in thoracic surgery. Severe postoperative pain may be encountered in patients undergoing VATS. Analgesic methods such as thoracic paravertebral block (TPVB), intercostal block and erector spina plane block (ESPB) are widely used for VATS. Among these methods, ultrasound (US) guided TPVB is the most preferred method. In recent years, the frequency of application of plane blocks as a component of multimodal analgesia has been increased. ESPB is one of them. Although there are publications showing that single-level ESPB applied from the T5 vertebra level spreads in the craniocaudal T3-L2 range, there are also publications stating that the spread is more limited. This study, it was aimed to compare the efficacy of bi-level ESPB application and one-level ESPB application for postoperative analgesia in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-40 kg/m2
* Patients undergoing elective video-assisted thoracoscopic surgery

Exclusion Criteria:

* Patient refusing the procedure
* History of chronic analgesic or opioid therapy
* History of local anesthetic allergy
* Infection in the intervention area
* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Pain scores | 1st hour after surgery
  Pain will be assessed at the first-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain scores | 2nd-hour after surgery.
  Pain will be assessed at the 2nd-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain scores | 4th-hour after surgery.
  Pain will be assessed at the 4th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain scores | 12th-hour after surgery.
  Pain will be assessed at the 12th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain scores | 24th-hour after surgery.
  Pain will be assessed at the 24th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain scores | 48th-hour after surgery.
  Pain will be assessed at the 48th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Postoperative intravenous morphine infusion therapy will be administered with the patient-controlled analgesia (PCA) method. Thanks to PCA, how much morphine the patient needs will be followed in mg.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Çankaya, Ankara
  - Ankara Atatürk Chest Diseases and Thoracic Surgery Training and Research Hospital, Keçiören, Ankara

REFERENCES:
- [Derived] Zengin EN, Yigit H, Cobas M, Salman N, Asli Demir Z. The analgesic effects of combined bilateral parasternal block and serratus anterior plane block for coronary artery bypass grafting surgery. BMC Anesthesiol. 2024 Aug 5;24(1):274. doi: 10.1186/s12871-024-02659-7. PMID 39103782
- [Derived] Zengin EN, Zengin M, Yigit H, Sazak H, Sekerci S, Alagoz A. Comparison of the effects of one-level and bi-level pre-incisional erector spinae plane block on postoperative acute pain in video-assisted thoracoscopic surgery; a prospective, randomized, double-blind trial. BMC Anesthesiol. 2023 Aug 11;23(1):270. doi: 10.1186/s12871-023-02232-8. PMID 37568076